CLINICAL TRIAL: NCT02505425
Title: Randomized Trial of ENABLE CHF-PC for Heart Failure Patients and Caregivers. (Comprehensive Heartcare For Patients and Caregivers)
Brief Title: ENABLE CHF-PC (Comprehensive Heartcare For Patients and Caregivers)
Acronym: ENABLE CHF PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Marie Anne Bakitas, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X140813007
Record Dates: First submitted 2015-07-08; First posted 2015-07-22 (Estimated); Results first posted 2021-02-11 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Intervention (Experimental): Behavioral: behavioral support
  Usual HF Care + ENABLE CHF-PC
  Interventions: Behavioral: Behavioral Support
- Usual HF Care (Active Comparator): Usual heart failure care includes any available supportive care resources and heart failure patient medical management based on national HF guidelines.
  Interventions: Behavioral: Usual HF Care

INTERVENTIONS:
Behavioral: Behavioral Support — ENABLE CHF-PC includes:
  1. In-person comprehensive Palliative Care Team (PCT) Consultation- as soon as feasible after enrollment.
  2. Palliative Care Nurse Coach (PNC) embedded within HF teams, instituting a phone-based 6-session patient and a 4-session caregiver curriculum followed by monthly phone-based supportive care for 48 weeks or patient death.
  The PNC uses the manualized curriculum: "Charting Your Course (CYC): An Intervention for Patients with Heart Failure and their Families".
  Usual Care: Usual heart failure care includes any available supportive care resources and heart failure patient medical management based on national HF guidelines.
  Other Names: ENABLE CHF-PC
  Arms: Active Intervention
Behavioral: Usual HF Care — Usual heart failure care includes any available supportive care resources and heart failure patient medical management based on national HF guidelines.
  Other Names: Usual Heart Failure Care
  Arms: Usual HF Care

SUMMARY:
Advanced heart failure affects nearly 6 million Americans, and less is known about how this illness affects the 80% of heart failure patients who are 65 years and older because research tends to focus on younger patients. Older patients with heart failure and their family caregivers, rarely have access to palliative supportive care services because the disease is unpredictable and palliative treatment may not be provided until after other medical treatments have been tried. Investigators are studying whether palliative care provided when advanced heart failure patients are still well will result in better quality of life, mood and less symptom distress compared to usual or standard heart failure care.

Specific Aims and Hypotheses:

Specific Aim 1: Determine whether ENABLE CHF-PC leads to higher advanced heart failure patient-reported quality of life (QOL) and mood (depression/anxiety); and lower symptom burden and resource use (e.g. hospital admissions and days, emergency visits) through 16 weeks post baseline.

• Hypothesis 1: Intervention participants will experience higher QOL and mood, and lower symptom burden and resource use through 16 weeks post baseline compared with those receiving usual HF care.

Specific Aim 2: Determine whether ENABLE CHF-PC leads to higher caregiver-reported QOL, mood (anxiety/depression), and self-reported health and lower caregiver burden through 16 weeks post baseline.

• Hypothesis 2: Intervention caregivers will report higher QOL, mood, and self-reported health, and lower caregiver burden through 16 weeks post baseline.

DETAILED DESCRIPTION:
As described.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read and understand English
2. NYHF III/IV heart failure (physician-determined)

Exclusion Criteria:

1. Dementia or significant confusion (Callahan 6-Item Cognitive Screening score ≤ 3)
2. DSM-IV Axis I diagnosis (e.g. schizophrenia, bipolar disorder, or active substance use disorder)
3. Patients will not be excluded if they do not identify a caregiver
4. Uncorrectable hearing loss.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 573 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2019-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bakitas, DNSc, Principal Investigator — University of Alabama at Birmimgham, School of Nursing, Dept. Acute, Chronic & Continuing Care
Locations (2):
- United States (2):
  - Birmingham Veterans Affairs Medical Center (BVAMC), Birmingham, Alabama
  - University of Alabama at Birmingham, School of Nursing, Dept. Acute, Chronic and Continuing Care, Birmingham, Alabama

IPD SHARING:
Plan to Share IPD: No
At this time, the study plans to share data in aggregate and as overall results only.

REFERENCES:
- [Derived] Wells R, Dionne-Odom JN, Azuero A, Buck H, Ejem D, Burgio KL, Stockdill ML, Tucker R, Pamboukian SV, Tallaj J, Engler S, Keebler K, Tims S, Durant R, Swetz KM, Bakitas M. Examining Adherence and Dose Effect of an Early Palliative Care Intervention for Advanced Heart Failure Patients. J Pain Symptom Manage. 2021 Sep;62(3):471-481. doi: 10.1016/j.jpainsymman.2021.01.136. Epub 2021 Feb 5. PMID 33556493
- [Derived] Stockdill ML, Dionne-Odom JN, Wells R, Ejem D, Azuero A, Keebler K, Sockwell E, Tims S, Burgio KL, Engler S, Durant R, Pamboukian SV, Tallaj J, Swetz KM, Kvale E, Tucker R, Bakitas M. African American Recruitment in Early Heart Failure Palliative Care Trials: Outcomes and Comparison With the ENABLE CHF-PC Randomized Trial. J Palliat Care. 2023 Jan;38(1):52-61. doi: 10.1177/0825859720975978. Epub 2020 Dec 1. PMID 33258422
- [Derived] Bakitas MA, Dionne-Odom JN, Ejem DB, Wells R, Azuero A, Stockdill ML, Keebler K, Sockwell E, Tims S, Engler S, Steinhauser K, Kvale E, Durant RW, Tucker RO, Burgio KL, Tallaj J, Swetz KM, Pamboukian SV. Effect of an Early Palliative Care Telehealth Intervention vs Usual Care on Patients With Heart Failure: The ENABLE CHF-PC Randomized Clinical Trial. JAMA Intern Med. 2020 Sep 1;180(9):1203-1213. doi: 10.1001/jamainternmed.2020.2861. PMID 32730613
- [Derived] Dionne-Odom JN, Ejem DB, Wells R, Azuero A, Stockdill ML, Keebler K, Sockwell E, Tims S, Engler S, Kvale E, Durant RW, Tucker RO, Burgio KL, Tallaj J, Pamboukian SV, Swetz KM, Bakitas MA. Effects of a Telehealth Early Palliative Care Intervention for Family Caregivers of Persons With Advanced Heart Failure: The ENABLE CHF-PC Randomized Clinical Trial. JAMA Netw Open. 2020 Apr 1;3(4):e202583. doi: 10.1001/jamanetworkopen.2020.2583. PMID 32282044
- [Derived] Wells R, Stockdill ML, Dionne-Odom JN, Ejem D, Burgio KL, Durant RW, Engler S, Azuero A, Pamboukian SV, Tallaj J, Swetz KM, Kvale E, Tucker RO, Bakitas M. Educate, Nurture, Advise, Before Life Ends Comprehensive Heartcare for Patients and Caregivers (ENABLE CHF-PC): study protocol for a randomized controlled trial. Trials. 2018 Aug 6;19(1):422. doi: 10.1186/s13063-018-2770-9. PMID 30081933

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruitment period was from October 2015 thru October 2018. Recruitment occurred at two sites: the University of Alabama at Birmingham (UAB) and the Birmingham Veterans Affairs Medical Center (BVAMC).
Groups:
- Active Intervention for Patients; Active Intervention for Caregivers: Behavioral: behavioral support
  Usual HF Care + ENABLE CHF-PC
  Behavioral Support: ENABLE CHF-PC includes:
  1. In-person comprehensive Palliative Care Team (PCT) Consultation- as soon as feasible after enrollment.
  2. Palliative Care Nurse Coach (PNC) embedded within HF teams, instituting a phone-based 6-session patient and a 4-session caregiver curriculum followed by monthly phone-based supportive care for 48 weeks or patient death.
  The PNC uses the manualized curriculum: "Charting Your Course (CYC): An Intervention for Patients with Heart Failure and their Families".
  Usual Care: Usual heart failure care includes any available supportive care resources and heart failure patient medical management based on national HF guidelines.
- Usual HF Care for Patients; Usual HF Care for Caregivers: Usual heart failure care includes any available supportive care resources and heart failure patient medical management based on national HF guidelines.
  Usual HF Care: Usual heart failure care includes any available supportive care resources and heart failure patient medical management based on national HF guidelines.
Period: Overall Study
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Started | 208 | 207 | 82 | 76
Completed | 120 | 125 | 32 | 50
Not Completed | 88 | 82 | 50 | 26
Not completed — Lost to Follow-up | 41 | 61 | 31 | 19
Not completed — Withdrawal by Subject | 39 | 9 | 19 | 7
Not completed — Death | 8 | 12 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers | Total
Number analyzed (Participants) | 208 | 207 | 82 | 76 | 573
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (8.0) | 64.1 (9.1) | 58.2 (12.4) | 57.6 (10.8) | 60.85 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 97 | 73 | 62 | 329
  Male | 111 | 110 | 9 | 14 | 244
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 113 | 113 | 46 | 36 | 308
  White | 92 | 92 | 32 | 38 | 254
  More than one race | 3 | 2 | 3 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants] — Southeast Region - AL, GA, MS, TN, FL
  Participants
    United States | 208 | 207 | 82 | 76 | 573

OUTCOME MEASURES:

1. Primary Outcome: Patient Quality of Life as Measured on the Kansas City Cardiomyopathy Questionnaire (KCCQ) Clinical Summary Score
Description: Baseline patient-reported Quality of Life (QOL) was measured on the Kansas City Cardiomyopathy Questionnaire (KCCQ) Clinical Summary Score, a heart failure-specific 23-item instrument. The KCCQ consists of 4 clinical domains: symptoms - frequency & severity; Physical Limitation; Quality of Life and Social Limitation and captures the patient's perspective of heart failure. Clinical summary scores range from 0 to 100. Higher KCCQ scores indicate better perceived health status. KCCQ clinical summary scores greater than or equal to 50 indicate good QOL.
Time Frame: Baseline
Population: This measure pertains to Patient Quality of Life (QOL). Caregiver QOL was analyzed using a different measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 208 | 207 | 0 | 0
score on a scale | 54.2 (20.5) | 51.1 (21.5) |  |

2. Primary Outcome: Patient Quality of Life as Measured on the Kansas City Cardiomyopathy Questionnaire (KCCQ) Clinical Summary Score
Description: Patient-reported Quality of Life (QOL) was measured on the Kansas City Cardiomyopathy Questionnaire (KCCQ) at 16 weeks. The KCCQ consists of 4 clinical domains: symptoms - frequency & severity; Physical Limitation; Quality of Life and Social Limitation and captures the patient's perspective of heart failure. Clinical summary scores range from 0 to 100. Higher KCCQ scores indicate better perceived health status. KCCQ clinical summary scores greater than or equal to 50 indicate good QOL.
Time Frame: 16 weeks
Population: This measure pertains to Patient Quality of Life (QOL) using the KCCQ. Caregiver QOL was analyzed using a different measure.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 120 | 125 | 0 | 0
score on a scale | 59.7 (1.8) | 54.8 (1.8) |  |

3. Primary Outcome: Patient Quality of Life as Measured on the Functional Assessment of Chronic Illness Therapy-Palliative Care Scale (FACIT-PAL-14)
Description: Baseline patient-reported Quality of Life (QOL) was measured on the Functional Assessment of Chronic Illness Therapy-Palliative Care Scale (FACIT-PAL-14). Scores range from 0 to 56; higher scores indicate better quality of life.
Time Frame: Baseline
Population: This measure pertains to Patient Quality of Life (QOL). Caregiver QOL was analyzed using a different measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 208 | 207 | 0 | 0
score on a scale | 36.8 (9.3) | 36.1 (9.7) |  |

4. Primary Outcome: Patient Quality of Life as Measured on the Functional Assessment of Chronic Illness Therapy-Palliative Care Scale (FACIT-PAL-14)
Description: Patient-reported Quality of Life (QOL) was measured on the Functional Assessment of Chronic Illness Therapy-Palliative Care Scale (FACIT-PAL-14) at 16 weeks. Scores range from 0 to 56; higher scores indicate better quality of life.
Time Frame: 16 weeks
Population: This measure pertains to Patient Quality of Life (QOL). Caregiver QOL was analyzed using a different measure. One intervention participant and two usual care participants did not provide sufficient responses to contribute to this outcomes measure score at 16 weeks.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 119 | 123 | 0 | 0
score on a scale | 38.5 (0.8) | 36.8 (0.8) |  |

5. Primary Outcome: Patient & Caregiver Mood - Anxiety - as Measured on the Hospital Anxiety and Depression Scale (HADS)
Description: Baseline patient & caregiver-reported mood - Anxiety - was measured on the Hospital Anxiety and Depression Scale (HADS). 7 items measure anxiety symptoms.Scores range from 0 to 21; higher scores indicate more severe symptoms.
Time Frame: Baseline
Population: This measure pertains to Patient & Caregiver Mood - Anxiety HADS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 208 | 207 | 82 | 76
score on a scale | 6.6 (3.5) | 6.8 (3.7) | 3.9 (3.1) | 3.7 (2.9)

6. Primary Outcome: Patient & Caregiver Mood - Anxiety - as Measured on the Hospital Anxiety and Depression Scale (HADS)
Description: Change from baseline in patient & caregiver-reported mood - Anxiety was measured on the HADS. 7 items measure anxiety symptoms. Scores range from 0 to 21; higher scores indicate more severe symptoms.
Time Frame: 16 weeks
Population: This measure pertains to Patient & Caregiver Mood - Anxiety HADS. One intervention patient and three usual care patients did not provide sufficient responses to contribute to this outcomes measure score at 16 weeks.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 119 | 122 | 32 | 50
score on a scale | 6.6 (0.3) | 7.1 (0.3) | 3.8 (0.5) | 4.2 (0.4)

7. Primary Outcome: Patient & Caregiver Mood - Depression - as Measured on the Hospital Anxiety and Depression Scale (HADS)
Description: Baseline patient and caregiver-reported depression was measured on the Hospital Anxiety and Depression Scale (HADS). 7 items measure depression symptoms. Scores range from 0 to 21; higher scores indicate more severe symptoms.
Time Frame: Baseline
Population: This measure pertains to Patient and Caregiver Mood - Depression Scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 208 | 207 | 82 | 76
score on a scale | 5.7 (4.3) | 5.8 (4.2) | 4.7 (3.1) | 4.8 (3.3)

8. Primary Outcome: Patient & Caregiver Mood - Depression - as Measured on the Hospital Anxiety and Depression Scale (HADS)
Description: Patient and caregiver-reported depression was measured on the Hospital Anxiety and Depression Scale (HADS) at 16 weeks. 7 items measure depression symptoms. Scores range from 0 to 21; higher scores indicate more severe symptoms.
Time Frame: 16 weeks
Population: This measure pertains to Patient and Caregiver Mood - Depression Scale. One intervention patient and three usual care patients did not provide sufficient responses to contribute to this outcomes measure score at 16 weeks.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 119 | 122 | 32 | 50
score on a scale | 4.9 (0.3) | 5.6 (0.3) | 4.5 (0.5) | 4.4 (0.4)

9. Primary Outcome: Caregiver Quality of Life as Measured on the Bakas Caregiving Outcomes Scale (BCOS)
Description: Baseline caregiver-reported quality of life (QOL) was measured on the Bakas Caregiving Outcomes Scale (BCOS). Score range: 15-105; higher scores indicate higher quality of life.
Time Frame: Baseline
Population: This measure was conducted among Caregiver participants only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 0 | 0 | 82 | 76
score on a scale |  |  | 65.0 (12.9) | 60.7 (10.4)

10. Primary Outcome: Caregiver Quality of Life as Measured on the Bakas Caregiving Outcomes Scale (BCOS)
Description: Caregiver-reported quality of life (QOL) was measured on the Bakas Caregiving Outcomes Scale (BCOS) at 16 weeks. Score range: 15-105; higher scores indicate higher quality of life.
Time Frame: 16 weeks
Population: This measure conducted among Caregiver participants only.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 0 | 0 | 32 | 50
score on a scale |  |  | 66.9 (2.1) | 63.9 (1.7)

11. Primary Outcome: Caregiver Burden - Objective - as Measured on the Montgomery Borgatta Caregiver Burden Scale (MBCB)
Description: Baseline caregiver-reported Objective burden was measured on the Montgomery Borgatta Caregiver Burden Scale (MBCB). This subscale measures the object burden, interference with the caregiver's day-to-day activities given caregiving demands. Score range: 6-30, Greater than 23 indicates high burden.
Time Frame: Baseline
Population: Montgomery Borgatta Caregiver Burden Scale (MBCB) was measured among Caregivers only.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 0 | 0 | 82 | 76
score on a scale |  |  | 20.1 (2.8) | 20.0 (2.9)

12. Primary Outcome: Caregiver Burden - Objective - as Measured on the Montgomery Borgatta Caregiver Burden Scale (MBCB)
Description: Caregiver-reported Objective burden was measured on the Montgomery Borgatta Caregiver Burden Scale (MBCB) at 16 weeks. This subscale measures the object burden, interference with the caregiver's day-to-day activities given caregiving demands.Score range: 6-30, Greater than 23 indicates high burden.
Time Frame: 16 weeks
Population: Montgomery Borgatta Caregiver Burden Scale (MBCB) was measured among Caregivers only.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 0 | 0 | 32 | 50
score on a scale |  |  | 20.2 (0.5) | 19.7 (0.4)

13. Primary Outcome: Caregiver Burden - Demand - as Measured on the Montgomery Borgatta Caregiver Burden Scale (MBCB)
Description: Baseline caregiver-reported Demand burden was measured on the Montgomery Borgatta Caregiver Burden Scale (MBCB). This subscale measures the demand burden or the strain among caregivers from meeting the needs of the care recipient. Score range: 6-30, Greater than 23 indicates high burden.
Time Frame: Baseline
Population: Montgomery Borgatta Caregiver Burden Scale (MBCB) was measured among Caregivers only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 0 | 0 | 82 | 76
score on a scale |  |  | 11.6 (2.5) | 11.6 (1.8)

14. Primary Outcome: Caregiver Burden - Demand - as Measured on the Montgomery Borgatta Caregiver Burden Scale (MBCB)
Description: Caregiver-reported Demand burden was measured on the Montgomery Borgatta Caregiver Burden Scale (MBCB) at 16 weeks. This subscale measures the demand burden or the strain among caregivers from meeting the needs of the care recipient. Score range: 6-30, Greater than 23 indicates high burden.
Time Frame: 16 weeks
Population: Montgomery Borgatta Caregiver Burden Scale (MBCB) was measured among Caregivers only.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 0 | 0 | 32 | 50
score on a scale |  |  | 11.1 (0.4) | 11.6 (0.3)

15. Primary Outcome: Caregiver Burden - Stress - as Measured on the Montgomery Borgatta Caregiver Burden Scale (MBCB)
Description: Baseline caregiver-reported Stress burden was measured on the Montgomery Borgatta Caregiver Burden Scale (MBCB). his subscale indicates the stress burden or emotional stress from the demands of caregiving. Score range: 6-30, Greater than 23 indicates high burden.
Time Frame: Baseline
Population: Montgomery Borgatta Caregiver Burden Scale (MBCB) was conducted among Caregivers only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 0 | 0 | 82 | 76
score on a scale |  |  | 12.3 (2.4) | 12.3 (2.2)

16. Primary Outcome: Caregiver Burden - Stress- as Measured on the Montgomery Borgatta Caregiver Burden Scale (MBCB)
Description: Caregiver-reported Stress burden was measured on the Montgomery Borgatta Caregiver Burden Scale (MBCB) at 16 weeks. This subscale indicates the stress burden or emotional stress from the demands of caregiving. Score range: 6-30, Greater than 23 indicates high burden.
Time Frame: 16 weeks
Population: Montgomery Borgatta Caregiver Burden Scale (MBCB) was measured among Caregivers only.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 0 | 0 | 32 | 50
score on a scale |  |  | 11.7 (0.4) | 12.2 (0.3)

17. Secondary Outcome: Patient and Caregiver PHYSICAL Health Status as Measured on the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form Global Health-10
Description: Baseline patient- and caregiver-reported PHYSICAL health status was measured on the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form Global Health-10. The PROMIS SF Global Health-10 measures general domains of health including physical, mental, and social health, symptoms, overall quality of life. Summed scores for PROMIS measures are converted to T scores with a mean of 50 and standard deviation of 10 in the general US population; higher scores indicate better functioning.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 208 | 207 | 82 | 76
score on a scale | 38.6 (8.0) | 38.1 (8.0) | 46.9 (8.9) | 48.0 (8.6)

18. Secondary Outcome: Patient and Caregiver PHYSICAL Health Status as Measured on the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form Global Health-10
Description: Patient- and caregiver-reported PHYSICAL health status was measured on the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form Global Health at 16 weeks. The PROMIS SF Global Health-10 measures general domains of health including physical, mental, and social health, symptoms, overall quality of life. Summed scores for PROMIS measures are converted to T scores with a mean of 50 and standard deviation of 10 in the general US population; higher scores indicate better functioning.
Time Frame: 16 weeks
Population: One intervention and three usual care patients did not provide sufficient responses to contribute to this outcomes measure score at 16 weeks. One intervention patient and three usual care patients did not provide sufficient responses to contribute to this outcomes measure score at 16 weeks.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 119 | 122 | 32 | 50
score on a scale | 39.4 (0.7) | 38.8 (0.7) | 46.9 (8.9) | 48.0 (8.6)

19. Secondary Outcome: Patient and Caregiver MENTAL Health Status as Measured on the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form Global Health-10
Description: Baseline patient- and caregiver-reported MENTAL health status was measured on the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form Global Health. The PROMIS SF Global Health-10 measures general domains of health including physical, mental, and social health, symptoms, overall quality of life. Summed scores for PROMIS measures are converted to T scores with a mean of 50 and standard deviation of 10 in the general US population; higher scores indicate better functioning.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 208 | 207 | 82 | 76
score on a scale | 45.8 (8.6) | 44.9 (8.7) | 48.5 (7.1) | 48.1 (7.9)

20. Secondary Outcome: Patient and Caregiver MENTAL Health Status as Measured on the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form Global Health-10
Description: Patient- and caregiver-reported MENTAL health status was measured on the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form Global Health at 16 weeks. The PROMIS SF Global Health-10 measures general domains of health including physical, mental, and social health, symptoms, overall quality of life. Summed scores for PROMIS measures are converted to T scores with a mean of 50 and standard deviation of 10 in the general US population; higher scores indicate better functioning.
Time Frame: 16 weeks
Population: One intervention patient and three usual care patients did not provide sufficient responses to contribute to this outcomes measure score at 16 weeks.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 119 | 122 | 32 | 50
score on a scale | 45.9 (0.7) | 44.7 (0.7) | 47.7 (1.0) | 48.2 (0.9)

21. Secondary Outcome: Patient Symptom Burden as Measured on the Kansas City Cardiomyopathy Questionnaire (KCCQ) Symptom Items
Description: Baseline patient-reported symptom burden was measured on symptom-based items from the Kansas City Cardiomyopathy Questionnaire (KCCQ). Higher KCCQ scores indicate better perceived health status. The KCCQ Symptom burden domain consists of 8 items and quantifies the frequency, severity and change over time with clinical symptoms in heart failure, including fatigue, shortness of breath, paroxysmal nocturnal dyspnea and patients' edema/swelling. KCCQ symptom domain scores range from 0 to 100; A score of 50 is the threshold between unstable heart failure symptoms (<50) or stable heart failure symptoms (>=50).
Time Frame: Baseline
Population: This outcomes measure pertains to patient-reported symptom burden.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 208 | 207 | 0 | 0
score on a scale | 52.2 (22.1) | 50.9 (24.2) |  |

22. Secondary Outcome: Patient Symptom Burden Items as Measured on the Kansas City Cardiomyopathy Questionnaire (KCCQ) Symptom Items.
Description: Patient-reported symptom burden was measured on symptom-based items from the Kansas City Cardiomyopathy Questionnaire (KCCQ) at 16 weeks. Higher KCCQ scores indicate better perceived health status. The KCCQ Symptom burden domain consists of 8 items and quantifies the frequency, severity and change over time for clinical symptoms in heart failure, including fatigue, shortness of breath, paroxysmal nocturnal dyspnea and patients' edema/swelling. KCCQ symptom domain scores range from 0 to 100; A score of 50 is the threshold between unstable heart failure symptoms (<50) or stable heart failure symptoms (>=50).
Time Frame: 16 weeks
Population: This outcomes measure pertains to patient-reported symptom burden.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 120 | 125 | 0 | 0
score on a scale | 59.6 (2.0) | 55.3 (1.9) |  |

23. Secondary Outcome: Patient Pain Intensity as Measured on the Patient-Reported Outcomes Measurement Information System (PROMIS) 3-item Pain Intensity Scale
Description: Baseline patient-reported PAIN INTENSITY was measured on the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Scale. Higher pain scores indicate more pain. Score range: 0-100; Scores greater than 50 indicate high pain.
Time Frame: Baseline
Population: Measure conducted among patients only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 208 | 207 | 0 | 0
score on a scale | 46.8 (10.8) | 45.1 (10.5) |  |

24. Secondary Outcome: Patient Pain Intensity as Measured on the Patient-Reported Outcomes Measurement Information System (PROMIS) 3-item Pain Intensity Scale
Description: Patient-reported PAIN INTENSITY was measured on the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Scale at 16 weeks. Higher pain scores indicate more pain. Score range: 0-100; Scores greater than 50 indicate high pain.
Time Frame: 16 weeks
Population: Measure conducted among patients only. One intervention participant and three usual care participants did not provide sufficient responses to contribute to this outcomes measure score at 16 weeks.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 119 | 122 | 0 | 0
score on a scale | 45.8 (0.9) | 47.4 (0.9) |  |

25. Secondary Outcome: Patient Pain Interference as Measured on the Patient-Reported Outcomes Measurement Information System (PROMIS) 2-item Pain Interference Scale
Description: Baseline patient-reported PAIN INTERFERENCE was measured on the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Scale. Higher pain interference scores indicate more interference in daily life. Score range: 0-100; Scores greater than 50 indicate high pain.
Time Frame: Baseline
Population: This measure was conducted among patients only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 208 | 207 | 0 | 0
score on a scale | 55.4 (10.9) | 54.5 (10.7) |  |

26. Secondary Outcome: Patient Pain Interference as Measured on the Patient-Reported Outcomes Measurement Information System (PROMIS) 2-item Pain Interference Scale
Description: Patient-reported PAIN INTERFERENCE was measured on the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Scale at 16 weeks. Higher pain interference scores indicate more interference in daily life. Score range: 0-100; Scores greater than 50 indicate high pain.
Time Frame: 16 weeks
Population: Conducted among patients only. One intervention participant and three usual care participants did not provide sufficient responses to contribute to this outcomes measure score at 16 weeks.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 119 | 122 | 0 | 0
score on a scale | 54.3 (0.9) | 57.7 (0.9) |  |

27. Secondary Outcome: Patient Resource Use - Days in Hospital - as Measured on the Investigator-developed Instrument
Description: Baseline patient-reported health care utilization - Number of Days in Hospital, last two months - was measured on the Resource Use Questionnaire. This measure is an investigator-developed instrument to capture number of Inpatient days, ICU days, ED visits, hospice use, palliative care provider visits, AD completion, and DNR orders. The possible range of Days in Hospital is 0 Days to 60 Days (last/previous two months prior to this measure).
Time Frame: Baseline
Population: Patient resource use (e.g. hospital admissions and days, emergency visits) was only captured among patients.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 208 | 206 | 0 | 0
days | 2.59 [1.64 to 4.07] | 2.75 [1.74 to 4.34] |  |

28. Secondary Outcome: Patient Resource Use - Days in Hospital - as Measured on the Investigator-developed Instrument
Description: Patient-reported health care utilization - Number of Days in Hospital, last two months - was measured on the Resource Use Questionnaire at 16 weeks. This measure is an investigator-developed instrument to capture number of Inpatient days, ICU days, ED visits, hospice use, palliative care provider visits, AD completion, and DNR orders. The possible range of Days in Hospital is 0 Days to 60 Days (last/previous two months prior to this measure).
Time Frame: 16 weeks
Population: Patient resource use (e.g. hospital admissions and days, emergency visits) was only captured among patients. One intervention participant and one usual care participant did not provide sufficient responses to contribute to this outcomes measure at 16 weeks.
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 119 | 124 | 0 | 0
days | 1.51 [0.82 to 2.77] | 1.29 [0.71 to 2.38] |  |

29. Secondary Outcome: Patient Resource Use - Emergency Department Visits - as Measured on the Investigator-developed Instrument
Description: Baseline patient-reported health care utilization - Number of Emergency Department Visits, last two months - was measured on the Resource Use Questionnaire. This measure is an investigator-developed instrument to capture number of Inpatient days, ICU days, ED visits, hospice use, palliative care provider visits, AD completion, and DNR orders. The possible range of Visits to ED is 0 Visits to 60 Visits (in the last/previous two months prior to this measure).
Time Frame: Baseline
Population: Patient resource use (e.g. hospital admissions and days, emergency visits) was only captured among patients. One participant in the Usual Care group did not respond to this survey item.
Measure: Mean (95% Confidence Interval); unit: visits
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 208 | 206 | 0 | 0
visits | 0.3 [0.23 to 0.4] | 0.28 [0.21 to 0.37] |  |

30. Secondary Outcome: Patient Resource Use - Emergency Department Visits - as Measured on the Investigator-developed Instrument
Description: Patient-reported health care utilization - Number of Emergency Department Visits, last two months - was measured on the Resource Use Questionnaire at 16 weeks. This measure is an investigator-developed instrument to capture number of Inpatient days, ICU days, ED visits, hospice use, palliative care provider visits, AD completion, and DNR orders. The possible range of Visits to ED is 0 Visits to 60 Visits (in the last/previous two months prior to this measure).
Time Frame: 16 weeks
Population: Patient resource use (e.g. hospital admissions and days, emergency visits) was only captured among patients. One intervention participant did not provide sufficient responses to contribute to this outcomes measure score at 16 weeks.
Measure: Mean (95% Confidence Interval); unit: visits
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
Number analyzed (Participants) | 119 | 125 | 0 | 0
visits | 0.17 [0.11 to 1.26] | 0.19 [0.13 to 0.28] |  |

ADVERSE EVENTS:
Time Frame: Baseline through 41 months
Description: All cause mortality: Patients - 41 were lost to follow-up & 39 withdrew among 208 patients enrolled and allocated to the intervention group; 61 were lost to follow-up & 9 withdrew of the 207 patients enrolled and allocated to the usual care group.
  Caregivers - 31 were lost to follow-up & 19 withdrew of the 82 caregivers enrolled and allocated to the intervention group; 19 were lost to follow-up & 7 withdrew of the 76 caregivers enrolled and allocated to the usual care group.
Arm/Group | Active Intervention for Patients | Usual HF Care for Patients | Active Intervention for Caregivers | Usual HF Care for Caregivers
All-Cause Mortality (participants affected / at risk) | 8/208 | 12/207 | 0/82 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/208 | 0/207 | 0/82 | 0/76
Other Adverse Events (participants affected / at risk) | 0/208 | 0/207 | 0/82 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/25/NCT02505425/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT02505425/ICF_001.pdf